CLINICAL TRIAL: NCT00051090
Title: Multicenter, Pilot Study of Telbivudine (LdT) Anti-HBV Treatment Prior to the Initiation of Highly Active Antiretroviral Therapy Containing Lamivudine in Subjects Coinfected With HBV and HIV
Brief Title: Treatment of Hepatitis B Virus (HBV) Before Beginning Anti-HIV Drugs in Patients With Both HBV and HIV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5167; 10962 (Registry Identifier: DAIDS ES); ACTG A5167
Record Dates: First submitted 2003-01-03; First posted 2003-01-06 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Hepatitis B
Keywords: Hepatitis B; Antiretroviral Therapy, Highly-Active; HIV Infections; Lamivudine; Reverse Transcriptase Inhibitors; Antiviral Agents; Drug Therapy, Combination; Treatment Naive
MeSH Terms: conditions — HIV Infections; Hepatitis B | interventions — Telbivudine; Lamivudine; efavirenz; Didanosine; abacavir

ARMS (1):
- A (Experimental): All eligible study participants
  Interventions: Drug: Telbivudine; Drug: Lamivudine; Drug: Efavirenz; Drug: Didanosine; Drug: Abacavir

INTERVENTIONS:
Drug: Telbivudine — Administered orally at a daily dosage of 600 mg for a period of 48 weeks
Drug: Lamivudine — Administered orally at a total daily dosage of 300 mg for Weeks 24-48
Drug: Efavirenz — Administered orally at a daily dose of 600 mg
Drug: Didanosine — Administered orally at a total dosage of either 400 mg or 250 mg determined by individual weight
Drug: Abacavir — Administered orally twice daily in doses of 300 mg

SUMMARY:
This study will evaluate the drug telbivudine (LdT) for treatment of hepatitis B virus (HBV) in HIV infected patients. Patients will take telbivudine alone for 24 weeks, add anti-HIV drugs for 24 weeks, then stop taking telbivudine while continuing their anti-HIV drug regimen. To enroll in this study, patients must not be taking any anti-HIV drugs and cannot have taken more than 31 days of treatment with lamivudine (3TC), protease inhibitors (PIs), or nonnucleoside reverse transcriptase inhibitors (NNRTIs).

DETAILED DESCRIPTION:
Studies indicate that 70% to 80% of HIV infected patients have or have had HBV infection and that 10% are HBV carriers. Lamivudine therapy for treatment of HBV in HIV infected patients has limited long-term efficacy due to the development of resistance mutations. Telbivudine is a thymidine analogue with excellent HBV inhibitory activity but no anti-HIV activity. The primary objective of this study is to evaluate the safety and anti-HBV activity of telbivudine alone and in combination with a lamivudine-based highly active antiretroviral therapy (HAART) regimen in patients coinfected with HBV and HIV.

Patients in this study will take telbivudine for 24 weeks. At Week 24, patients will add a HAART regimen containing lamivudine and efavirenz plus either didanosine or abacavir. Patients who are unable to add a HAART regimen at Week 24 due to lab abnormalities or other contraindications will be allowed to delay the initiation of HAART until Week 30. Patients may initiate HAART prior to Week 24 if deemed medically necessary by the primary HIV care provider. Patients will take both telbivudine and HAART for 24 weeks. At Week 48, patients will discontinue telbivudine and continue on the HAART regimen alone for an additional 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* No antiretroviral therapy within 6 months prior to study entry
* Less than 31 days cumulative therapy with lamivudine, a protease inhibitor, or a nonnucleoside reverse transcriptase inhibitor
* Willingness to delay HAART until at least Week 24 of study
* Ability to procure and initiate HAART regimen
* CD4+ cell count >= 250 cells/mm3 within 60 days prior to study entry
* HIV-1 RNA > 400 copies/ml within 60 days prior to study entry
* Serum HBV DNA >= 1,000,000 copies/ml within 60 days prior to study entry
* Positive serum hepatitis B surface antigen (HbsAG)
* Acceptable methods of contraception

Exclusion Criteria:

* Pregnancy or breast-feeding
* Allergy, sensitivity, or intolerance to study drugs
* Alcohol consumption averaging more than 1 drink/day within past 30 days
* Decompensated cirrhosis
* HCV antibody positive or known HCV RNA positive
* HDV antibody positive
* Certain medical conditions
* Use of certain medications with anti-HBV activity within 90 days of study entry
* Use of systemic corticosteroids within 30 days of study entry
* Use of any systemic antineoplastic, immunomodulatory treatment, or radiation within 24 weeks of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
HBV viral loads | At Study entry, Week 24 and Week 48
Safety and tolerability of telbivudine | Throughout study

SECONDARY OUTCOMES:
Safety and tolerability of HAART | Throughout study
Change in ALT level | Throughout study
HBV genetic mutation status at HBV virologic failure | Throughout study
HIV viral load | At Study entry, Weeks 24, 48, and 60
HBV viral load and hepatic transaminase concentrations | At Week 60

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Lynch, M.D., Study Chair — Northwestern University

REFERENCES:
- [Background] den Brinker M, Wit FW, Wertheim-van Dillen PM, Jurriaans S, Weel J, van Leeuwen R, Pakker NG, Reiss P, Danner SA, Weverling GJ, Lange JM. Hepatitis B and C virus co-infection and the risk for hepatotoxicity of highly active antiretroviral therapy in HIV-1 infection. AIDS. 2000 Dec 22;14(18):2895-902. doi: 10.1097/00002030-200012220-00011. PMID 11153671
- [Background] Sulkowski MS, Thomas DL, Chaisson RE, Moore RD. Hepatotoxicity associated with antiretroviral therapy in adults infected with human immunodeficiency virus and the role of hepatitis C or B virus infection. JAMA. 2000 Jan 5;283(1):74-80. doi: 10.1001/jama.283.1.74. PMID 10632283
- [Background] Sulkowski MS, Thomas DL, Mehta SH, Chaisson RE, Moore RD. Hepatotoxicity associated with nevirapine or efavirenz-containing antiretroviral therapy: role of hepatitis C and B infections. Hepatology. 2002 Jan;35(1):182-9. doi: 10.1053/jhep.2002.30319. PMID 11786975
- [Background] Benhamou Y, Bochet M, Thibault V, Di Martino V, Caumes E, Bricaire F, Opolon P, Katlama C, Poynard T. Long-term incidence of hepatitis B virus resistance to lamivudine in human immunodeficiency virus-infected patients. Hepatology. 1999 Nov;30(5):1302-6. doi: 10.1002/hep.510300525. PMID 10534354